CLINICAL TRIAL: NCT02699294
Title: Comparison of Effectiveness of Two Different Stretching Exercises Combined With Pressure Release Technique on Latent Trigger Points in The Pectoralis Minor Muscle
Brief Title: The Effect Of Stretching Exercise on Pectoralis Minor Myofascial Latent Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Research assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 34910702
Record Dates: First submitted 2015-11-16; First posted 2016-03-04 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Myofascial Trigger Point Pain
Keywords: Pain Threshold; Pectoralis Minor; Proprioceptive Neuromuscular Facilitation (PNF) Stretching; Physiotherapy; Rehabilitation
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Contract-relax PNF stretch (Experimental): A contract-relax PNF stretching techniques of the pectoralis minor muscle including latent trigger points will be applied by Group 1 after a single intervention of manual pressure release will be performed according to the techniques describe by Simons et al. (1999).
  Interventions: Other: Manual pressure release; Other: Contract-relax PNF stretch
- Z-stretch (Experimental): The Z- stretch of the pectoralis minor muscle including latent trigger points will be applied by Group 2 after a single intervention of manual pressure release will be performed according to the techniques describe by Simons et al. (1999).
  Interventions: Other: Manual pressure release; Other: Z-stretch
- Manual pressure release (Experimental): The single intervention of manual pressure release will be only applied to Group 3 according to the techniques describe by Simons et al. (1999).
  Interventions: Other: Manual pressure release
- Control (No Intervention): This is a control group.

INTERVENTIONS:
Other: Manual pressure release — Subjects will be positioned supine on a treatment plinth and will be encouraged to relax as much as possible before pressure is applied. A slow pressure to myofascial latent trigger point will be applied directly over the marked pectoralis minor muscle myofascial latent trigger point site until a moderate but tolerable pain value of 7 out of 10 (0= no pain, 10= severe pain) is reported. Constant pressure will be sustained for 90 seconds if the subjects report that the pain is decreased to a value of 3, the pressure will be increased to restore perceived pain to the value of 7. Then, tissue resistance (barrier) in pectoralis minor muscle will be controlled.
  Arms: Contract-relax PNF stretch; Manual pressure release; Z-stretch
Other: Contract-relax PNF stretch — Subjects will be in a sitting position with hands being clasped behind the head. The pectoralis minor muscle will be passively and slowly stretched until a strong but tolerable stretch discomfort intensity level of 4 out of 10 (0= no pain, 10= severe pain) is reported. Passive stretch will be sustained for 10 seconds followed by 6 seconds of maximal voluntary isometric contraction of the pectoralis minor muscle. Then, subjects will be instructed to relax for further 4 seconds. Subjects will maintain newly active stretched position of pectoralis minor muscle for 10 seconds with a strong but tolerable stretch discomfort intensity level of 4 out of 10. The procedure will be repeated four times with 30 seconds of rest between two successive trials.
  Arms: Contract-relax PNF stretch
Other: Z-stretch — Subjects will be positioned supine with knee bent on a treatment plinth, and the legs will be rotated to the opposite direction of the arm to be stretched placing a stabilizing distal tension on the ribs. Then, the subjects will be slowly brought the arm in a circular motion overhead pausing at the points of tightness, maintaining close contact to the treatment table until a strong but tolerable stretch discomfort intensity level of 4 out of 10 (0= no pain, 10= severe pain) is reported. Self-stretch of pectoralis minor muscle, including myofascial latent trigger points will be sustained for 30 seconds. The procedure will be repeated four times with 30 seconds of rest between two successive trials.
  Arms: Z-stretch

SUMMARY:
This randomised-controlled trial investigates whether a single intervention of manual pressure release combined with stretching exercise has an effect on muscle length, pain perception threshold, and respiratory function in subjects with latent myofascial trigger point in the pectoralis minor muscle or not. First quarter of the participants will receive a single intervention of manual pressure release combined with contract-relax PNF stretching exercise of pectoralis minor muscle, second quarter of the participants will receive a single intervention of manual pressure release combined with Z stretching exercise of pectoralis minor muscle while, only a single intervention of manual pressure release will be applied to third quarter of the participants and final quarter of them will not receive any intervention.

DETAILED DESCRIPTION:
Myofascial trigger points are hyperirritable points located within a taut band of skeletal muscle or fascia, which cause referred pain, local tenderness and autonomic changes when compressed. They are classified as either active myofascial trigger points (ATrPs) or latent myofascial trigger points (LTrPs). ATrPs can be inactivated by different treatment strategies; however, they never fully disappear but rather convert to the latent form. Therefore, the diagnosis and treatment of LTrPs is important. Invasive and noninvasive techniques are available for management of LTrPs. Invasive techniques include trigger point injections and dry needling whereas noninvasive techniques include manual therapy techniques and electrotherapy modalities. Manual therapy techniques for the treatment of myofascial trigger points include joint manipulation, strain/counterstrain, ischemic compression and pressure, massage therapy, myofascial release therapy, muscle energy techniques, point pressure release and transverse friction massage. Additionally, recent studies showed that the myofascial trigger point therapy combined with stretching exercise may be an effective for decreasing the pain level. However, there is insufficient evidence to determine what type stretching exercise is most effective and its immediate effects on muscle length in people with LTrPs. Therefore, the aim of this randomised-controlled trial is to investigate the effect on muscle length, pain perception threshold, and respiratory function after a single intervention of manual pressure release combined with stretching exercise on LTrPs in the pectoralis minor muscle.

The sample size and power calculations is performed with the sample size calculator (InStat). The calculations is based on a standard deviation of 0.5 points, the minimal clinically important difference (MCID) for Pectoralis Minor Index of 0.89 points, an alpha level of 0.05, a β level of 5%, and a desired power of 95%. These parameters generate a sample size of at least 9 participants for each group. Total of 40 subjects will be recruited into the study in order to allow for a loss to follow-up.

Potential participants will be invited through the posting of flyers at Istanbul University, Turkey. Flyer recruitment method will be used in this trial because it is the most effective, yielding the highest number of enrolments. All participants will be completed an informed consent form that described the purpose and procedures of testing. prior to participating in the study. Forty participants fitting the inclusion criteria will be randomly assigned to one of four parallel groups (ratio 1:1:1:1). For allocation of the participants, "Randomization.com" which is an online, randomisation web service will be used (http://www.randomization.com/). Simple randomisation procedures (computerized random numbers) will be done and sequentially numbered index cards with the random assignment will be prepared by an investigator with no clinical involvement in the study. The index cards will be folded and placed in sealed opaque envelopes. Then, the blind investigator will open each envelope and allocate the participants to group according to selected index card. The interventions will be performed by the same physiotherapist at a university research clinic, and assessments and data collection will be made by another therapist. Whereas interventionist will be aware of the allocated arm, patients and outcome assessor will be kept blind to allocation.

The data will be evaluated using the Statistical Package for the Social Sciences 21.0 program for Windows and by analyzing descriptive statistics (frequency, mean and standard deviation). Kolmogorov-Smirnov Test will be used to assess the distribution of data. The one-way analysis of variance (ANOVA) for repeated measures with the Bonferroni post hoc test will used to determine whether differences in the mean scores of outcome measure among three time points (baseline, immediate after and 24 hours later) between study groups. In this study, p values less than 0.05 will be regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with at least one latent myofascial trigger point in the pectoralis minor muscle

Exclusion Criteria:

* Presence of active trigger points in the pectoralis minor muscle
* Any orthopaedic problems pertaining to the spine-shoulder complex (e.g., fractures, arthrosis, listhesis, sprains, strains) within the last six months
* Surgery on the spine-shoulder complex before the study
* Neurological impairment in the upper extremities
* Receiving the treatment for myofascial pain within the last three months
* Receiving anti-inflammatory and pain relief medication in the past 24 hours

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pectoralis minor index (PMI) to 24 hours follow-up | Baseline, immediately after intervention, and 24 hours follow-up
  The PMI will be calculated by dividing the resting muscle length measurement by the subject height in centimeters and multiplying by 100. The test-retest reliability for PMI measurement is 0.94 (95 % Confidence Interval (CI): 0.81-0.98).

SECONDARY OUTCOMES:
Pectoralis minor length | Baseline, immediately after intervention, and 24 hours follow-up
  The resting length of the pectoralis minor can be validly measured using palpable landmarks and can be reliably measured with a caliper or a cloth tape measure. These landmarks are (1) the inferomedial aspect of the coracoid process and (2) the caudal edge of the fourth rib at the sternum. The distance in centimeters between these bony reference points will be measured with using a tape measure.
Pain pressure threshold of pectoralis minor muscle myofascial latent trigger point site | Baseline, immediately after intervention, and 24 hours follow-up
  Digital pressure algometry showed high intra-rater reliability for pressure pain threshold measurements which might be a useful parameter in assessing the effects of treatment for musculoskeletal pain and myofascial pain syndrome.
Rounded shoulder posture measure | Baseline, immediately after intervention, and 24 hours follow-up
  There is no significant difference between the concurrent validity of the supine rounded shoulder posture measure an a seated assessment of scapular posture. Rounded shoulder posture will be measured from the acromion to the wall behind the subject to determine the amount of forward displacement with using a levelled metric ruler
The Forced Vital Capacity (FVC) | Baseline and 24 hours follow-up
  The Forced Vital Capacity (FVC) (Liter (L) will be assessed by using a portable spirometer.
Forced Expiratory Volume in 1 second (FEV1) | Baseline and 24 hours follow-up
  Forced Expiratory Volume in 1 second (FEV1) (L) will be assessed by using a portable spirometer.
The FEV1/FVC ratio | Baseline and 24 hours follow-up
  The FEV1/FVC ratio (% of predicted normal) will be assessed by using a portable spirometer.
Peak Expiratory Flow (PEF) | Baseline and 24 hours follow-up
  Peak Expiratory Flow (PEF) (L/s) will be assessed by using a portable spirometer.
Maximum Inspiratory Pressure (MIP) | Baseline and 24 hours follow-up
  Maximum Inspiratory Pressure (MIP) will be assessed by using a hand-held respiratory pressure meter (cmH2O).
Maximal Expiratory Pressure (MEP) | Baseline and 24 hours follow-up
  Maximal Expiratory Pressure (MEP) will be assessed by using a hand-held respiratory pressure meter (cmH2O).

OTHER OUTCOMES:
Visual Analogue Scale (VAS) | Baseline
  The VAS is used for which a patient is asked to indicate his/her perceived pain during the rest and activity times. Respondents will mark the location on the 10-centimeter (cm) line corresponding to the amount of pain they experienced.
Disability arm shoulder hand questionnaire (DASH) | Baseline
  The DASH questionnaire is a region-specific, self-report scale to evaluate health status of upper extremity disabilities.
Short-Form 12 | Baseline
  The Short-Form 12 questionnaire is an instrument for evaluating health and quality of life perception.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PT, Principal Investigator — Research Assistant; Ebru Kaya Mutlu, PhD, PT, Study Director — Lecturer; Rustem Mustafaoglu, MSc, PT, Principal Investigator — Research Assistant; Arzu Razak Ozdincler, Prof. Dr, Study Chair — Professor
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trampas A, Kitsios A, Sykaras E, Symeonidis S, Lazarou L. Clinical massage and modified Proprioceptive Neuromuscular Facilitation stretching in males with latent myofascial trigger points. Phys Ther Sport. 2010 Aug;11(3):91-8. doi: 10.1016/j.ptsp.2010.02.003. Epub 2010 May 5. PMID 20673857
- [Background] Borstad JD. Measurement of pectoralis minor muscle length: validation and clinical application. J Orthop Sports Phys Ther. 2008 Apr;38(4):169-74. doi: 10.2519/jospt.2008.2723. Epub 2007 Nov 21. PMID 18434665
- [Background] Celik D, Mutlu EK. Clinical implication of latent myofascial trigger point. Curr Pain Headache Rep. 2013 Aug;17(8):353. doi: 10.1007/s11916-013-0353-8. PMID 23801006
- [Background] Halbertsma JP, van Bolhuis AI, Goeken LN. Sport stretching: effect on passive muscle stiffness of short hamstrings. Arch Phys Med Rehabil. 1996 Jul;77(7):688-92. doi: 10.1016/s0003-9993(96)90009-x. PMID 8669996
- [Background] Hanten WP, Olson SL, Butts NL, Nowicki AL. Effectiveness of a home program of ischemic pressure followed by sustained stretch for treatment of myofascial trigger points. Phys Ther. 2000 Oct;80(10):997-1003. PMID 11002435
- [Background] Borstad JD, Ludewig PM. Comparison of three stretches for the pectoralis minor muscle. J Shoulder Elbow Surg. 2006 May-Jun;15(3):324-30. doi: 10.1016/j.jse.2005.08.011. PMID 16679233
- [Background] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Background] Lee JH, Cynn HS, Yoon TL, Ko CH, Choi WJ, Choi SA, Choi BS. The effect of scapular posterior tilt exercise, pectoralis minor stretching, and shoulder brace on scapular alignment and muscles activity in subjects with round-shoulder posture. J Electromyogr Kinesiol. 2015 Feb;25(1):107-14. doi: 10.1016/j.jelekin.2014.10.010. Epub 2014 Oct 28. PMID 25467545
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Wong CK, Coleman D, diPersia V, Song J, Wright D. The effects of manual treatment on rounded-shoulder posture, and associated muscle strength. J Bodyw Mov Ther. 2010 Oct;14(4):326-33. doi: 10.1016/j.jbmt.2009.05.001. Epub 2009 Jun 26. PMID 20850039
- [Background] Carlsson AM. Assessment of chronic pain. I. Aspects of the reliability and validity of the visual analogue scale. Pain. 1983 May;16(1):87-101. doi: 10.1016/0304-3959(83)90088-X. PMID 6602967
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- See also: Simons et al., 1999 — https://books.google.com.tr/books?id=63OYdoNBNC8C&redir_esc=y